CLINICAL TRIAL: NCT04768543
Title: Stimulation Therapy for Apnea: Reporting Thoughts
Acronym: START
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Principal Investigator, Faith Luyster, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY20090150
Record Dates: First submitted 2021-02-16; First posted 2021-02-24 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; upper airway stimulation therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Exposure: Patients with moderate to severe OSA treated with UAS (Inspire Medical Systems, Inc)
  Interventions: Device: Upper airway stimulation (Inspire Medical Systems, Inc.)

INTERVENTIONS:
Device: Upper airway stimulation (Inspire Medical Systems, Inc.) — phasic hypoglossal nerve stimulation device

SUMMARY:
Upper airway stimulation (UAS) via unilateral implantation of a phasic hypoglossal nerve stimulation device is a safe and effective alternative treatment for patients with moderate to severe obstructive sleep apnea (OSA) who are unwilling or unable to adhere to positive airway pressure (PAP) therapy. Although adherence to UAS is higher than to PAP, there remain patients who are not using UAS consistently. The aim of this project is to explore critical factors in the use of UAS by OSA patients using qualitative research methods (personal interviews). The proposed study will provide crucial information about patients' concerns regarding UAS use and suggestions for how to support new UAS recipients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* ADHERE registry patient
* Received UAS implant from June 2017 to present

Exclusion Criteria:

* Patients without up to date contact information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe OSA treated with UAS (Inspire Medical Systems, Maple Grove, Minnesota) who are part of the ADHERE registry.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Experiences with UAS therapy | up to 4 years
  individual qualitative interview via telephone

CONTACTS AND LOCATIONS:
Overall Officials: Faith Luyster, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Luyster FS, Ni Q, Lee K, Harrison C, Ramprasad VH, Soose RJ, Strollo PJ. Factors affecting obstructive sleep apnea patients' use of upper airway stimulation treatment. J Clin Sleep Med. 2022 Sep 1;18(9):2207-2215. doi: 10.5664/jcsm.10086. PMID 35689597